CLINICAL TRIAL: NCT03827694
Title: Non-Invasive Diagnosis of Pediatric Pulmonary Invasive Mold Infections
Acronym: DOMINIC
Status: Recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Children's Hospital of Philadelphia (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00094558; R01AI139032 (NIH)
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Invasive Fungal Infections; Pulmonary Invasive Aspergillosis
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with possible PIFI
  Interventions: Diagnostic Test: Non-Invasive Testing for PIFI

INTERVENTIONS:
Diagnostic Test: Non-Invasive Testing for PIFI — galactomannan assay, fungal PCRs, cell-free next-generation DNA/RNA sequencing, RNAseq

SUMMARY:
This study will establish a non-invasive diagnostic approach and evaluate clinical outcomes for children at high-risk for pulmonary invasive fungal infection (PIFI).

ELIGIBILITY:
Inclusion Criteria:

* Males or females age > 120 days and < 22 years at any participating site
* Have at least one of the following conditions associated with a known high incidence of IFI: hematopoietic stem cell transplantation (HSCT), aplastic anemia, bone marrow failure, primary or acquired immune deficiency, or malignancy
* New (last 96 hours) radiographic evidence of at least one of the following: at least one nodular lesion greater than or equal to 5 mm in size, a wedge-shaped and segmental or lobar consolidation, a cavitary lesion, a lesion with a halo sign, a lesion with a reverse halo sign, or a lesion with an air crescent sign
* Prolonged neutropenia (absolute neutrophil count < 500 cells/µl for a period of ≥ 5 consecutive days) in 30 days prior to and including the day of qualifying chest MRI or CT scan date OR currently receiving systemic therapy for acute or chronic graft-versus-host disease (GVHD) OR presence of neutrophil dysfunction because of underlying acquired or primary immune deficiency (e.g. chronic granulomatous disease) on the date of the qualifying chest MRI or CT scan
* Subject consent or parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria:

* Weight <3 kg, so as to not exceed 3 ml/kg in a single blood draw
* Previous inclusion in this study

Ages: 120 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients receiving care at a participating study site
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Likelihood ratio of the galactomannan assay to return a positive result among subjects determined to have PIFI | Baseline
Likelihood ratio of galactomannan assay to return a negative result among subjects determined not to have PIFI | Baseline
Likelihood ratio of fungal PCRs (Aspergillus PCR, Mucorales PCR) to return a positive result among subjects determined to have PIFI | Baseline
Likelihood ratio of fungal PCRs (Aspergillus PCR, Mucorales PCR) to return a negative result among subjects determined not to have PIFI | Baseline
Likelihood ratio of cell-free next generation DNA/RNA sequencing identifying a fungal pathogen to return a positive result among subjects determined to have PIFI | Baseline
Likelihood ratio of cell-free next generation DNA/RNA sequencing identifying a fungal pathogen to return a negative result among subjects determined not to have PIFI | Baseline
Likelihood ratio of molecular RNAseq platform assessing host immune response to return a positive result among subjects determined to have PIFI | Baseline
Likelihood ratio of molecular RNAseq platform assessing host immune response to return a negative result among subjects determined not to have PIFI | Baseline

SECONDARY OUTCOMES:
Composite outcome score between patients with possible pulmonary invasive fungal infection managed with empirical antifungal therapy versus an invasive diagnostic procedure | 49 days
  Outcome score inclusive of outcomes and adverse events. Comprehensive clinical outcome score from most to least desirable are score of 1 (survival, improvement in pulmonary nodules, no adverse events related to anti-fungal therapy or invasive diagnostic intervention) to score of 7 (death)

CONTACTS AND LOCATIONS:
Overall Officials: William Steinbach, Principal Investigator — University of Arkansas; Brian Fisher, Principal Investigator — Children's Hospital of Philadelphia
Locations (33):
- United States (32):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - Rady Children's Hospital, UCSD, La Jolla, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital, Stanford University, Palo Alto, California
  - University of California San Francisco, Benioff Children's Hospital, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - All Children's Research Institute, St. Petersburg, Florida
  - Emory University-Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medicine, Comer Children's, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota
  - Children's Mercy, Kansas City, Missouri
  - The Washington University, St Louis, Missouri
  - Children's Omaha, Omaha, Nebraska
  - Weil Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Ascension Seton Medical Center, Austin, Texas
  - University of Texas Southwest Medical Center (UTSW), Dallas, Texas
  - MD Anderson, Houston, Texas
  - Seattle Children's Research Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada